CLINICAL TRIAL: NCT06038474
Title: Descartes-08 for Patients With Systemic Lupus Erythematosus
Acronym: SLE-001
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC08-SLE-001
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Descartes-08; CART; CAR-T; Autoimmune; Auto-antibody; Auto antibody; chimeric antigen receptor; T cells; Lupus; SLE; Lupus Erythematosus; Systemic Lupus Erythematosus; LE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Descartes-08 (Other): Drug: Descartes-08
  Autologous T-cells expressing a chimeric antigen receptor directed to BCMA
  Interventions: Drug: Descartes-08

INTERVENTIONS:
Drug: Descartes-08 — Autologous T-cells expressing a chimeric antigen receptor directed to BCMA

SUMMARY:
This is a Phase II study to evaluate the safety, tolerability and manufacturing feasibility of Descartes-08 CAR T-cells in patients with Systematic Lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age.
* Patient must have systemic lupus erythematosus (SLE) at the time of screening.
* Active symptoms despite recent or ongoing immunosuppressive therapy with glucocorticoids and at least 2 other immunosuppressive medications being tried for at least 12 weeks within 24 months of screening.
* At least one of: anti-dsDNA, anti-histone, anti-chromatin, and/or anti-Sm antibodies detectable at screening as assessed by a CLIA-certified laboratory.

Exclusion Criteria:

* Active severe lupus nephritis, active severe CNS lupus, and/or neurological symptoms of SLE including headache, seizure, psychosis, and organic brain syndrome (a patient with an incidental headache, deemed unrelated to SLE, may re-screen by telephone upon resolution of the headache);
* Major chronic illness that is not well managed at the time of study entry and in the opinion of the investigator may increase the risk to the patient.
* Patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Assess safety and tolerability of Descartes-08 in patients with systemic lupus erythematosus (SLE) | Day -59 to Day 50
  Results will be descriptive. Safety and tolerability endpoints will include descriptive statistics of AEs and SAEs. Patients must be followed until all AEs have resolved to Grade 2 or less except for lymphopenia and alopecia.

SECONDARY OUTCOMES:
Quantify the clinical activity of Descartes-08 in patients with SLE using Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | Day -59 to Month 12
  Assessment of Systemic Lupus Erythematosus Disease Activity Index 2000 from baseline administration at various timepoints up to month 12 follow up visit. A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
Assess the clinical activity of Descartes-08 in patients with SLE using Systemic Lupus Erythematosus Responder Index (SRI) | Day -59 to Month 12
  Assessment of whether participants meet the Systemic Lupus Erythematosus Responder Index (SRI) criteria (Yes/No) at various timepoints up to month 12 follow up visit.
Assess the clinical activity of Descartes-08 in patients with SLE using British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment (BICLA) | Day -59 to Month 12
  Assessment of whether participants meet the British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment (BICLA) criteria (Yes/No) at various timepoints up to month 12 follow up visit.
Quantify the clinical activity of Descartes-08 in patients with SLE using Physician Global Assessment (PGA) | Day -59 to Month 12
  Assessment of Physician Global Assessment (PGA) from baseline administration at various timepoints up to month 12 follow up visit. A total score can fall between 0.0 and 3.0, with a higher score representing a more significant degree of disease activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Profound Research LLC, Oceanside, California, United States

IPD SHARING:
Plan to Share IPD: No